CLINICAL TRIAL: NCT03280069
Title: Evaluation of Ocular Surface Changes Following RF Electrocoagulation Treatment of the Periorbital Region
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ophthalmic Consultants of Long Island (Other)
Responsible Party: Principal Investigator, Gerard D'Aversa, MD, Principal Investigator, Ophthalmic Consultants of Long Island
Other Study IDs: OCLI-RFE-10D
Record Dates: First submitted 2017-09-08; First posted 2017-09-12 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Skin Laxity; Meibomian Gland Dysfunction
MeSH Terms: conditions — Cutis Laxa; Meibomian Gland Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Subjects between the ages of 40 - 70: Subjects who present with signs of skin laxity & evaporation dry eye will receive 3 treatments with the THERMIeyes® 20 RF System and monitored for improvements in the conditions for which they have presented.
  Interventions: Device: THERMIeyes® 20 RF System

INTERVENTIONS:
Device: THERMIeyes® 20 RF System — The masked evaluating physician will be blinded as to which eye is treated. The evaluation on all visits will be performed on both eyes by the masked physician who will not know which eye has been treated with the THERMIeyes® 20 RF System. The treating technician will be aware of the treated eye so as to ensure all treatments are performed to the same eye.

SUMMARY:
This protocol will evaluate THERMIeyes® for its ability to treat periorbital skin laxity and wrinkles and monitor ocular surface changes and their effect on evaporative dry eye associated with MGD.

DETAILED DESCRIPTION:
Subjects with skin laxity and evaporative dry eye will be recruited for enrollment in this study. Subjects must present with subjective and objective indicators for periorbital skin laxity and wrinkle grade of 2 or greater out of a 4 point scale. To qualify, subjects must present with high symptoms score on subjective Ocular Surface Disease Index© (OSDI©) Questionnaires (scores≥ 15); Rapid Tear Break up (< 5 seconds) and Grade ≥ 1 of Flourescein Staining in one area of the cornea. Each of these parameters are to be assessed prior to treatment and at each follow up visit. Treatment is to be performed on periorbital skin only around one eye of the subject using the THERMIeyes® standard protocol. This may result in some redness of the periorbital skin. Subjects are to be seen and treated 2-3 weeks apart for a total of 3 treatments. Subjects will be followed at 6 and 12 weeks after the final treatment. A Validated Grading Scale for Crow's Feet will be used to evaluate changes in skin wrinkles and dry eye signs and symptoms scores will be compared with pre-treatment findings.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 40-70 Inclusive; Male or Female
* Subjects must demonstrate subjective and objective indicators for periorbital skin laxity and wrinkle grade of 2 or greater out of a 4 point scale
* Subjects must have an OSDI© score of ≥ 15,
* Subjects must have a Grade 1 or higher staining pattern with fluorescein stain in any area of the cornea.
* The subjects may continue their current treatment for dry eye including the use of artificial tears, gels or ointments. They are to continue any topical medications for dry eye such as Cyclosporin or Lifitegrast. Subjects may continue to take chronic medications systemically including anti-inflammatory medications (aspirin, NSAIDS, Prednisone) as long as the dose and frequency is not changed throughout the study.
* Subjects may be included if they have punctual plugs present in any tear duct. If a plug comes out during the study it may be re-inserted so that the Subject is returned to their pre-treatment baseline state.
* Women of childbearing years should have pregnancy testing performed to ensure that pregnancy has not occurred during the study. Urine pregnancy screening will be performed prior to any treatment and on follow up visits until the study is completed

Exclusion Criteria:

* The subject must meet the inclusion criteria as listed
* During the study they cannot have any new medications started that are anti-inflammatory in nature. This includes topical steroids, Lifitegrast, cyclosporine or systemic medications such as steroids, NSAIDS, aspirin, Doxycyline or other Macrolid antibiotics.
* Subjects cannot have a punctual plug inserted into a tear duct that has not had a plug present prior to the start of the study.
* Participation in other clinical trials during the course of this study is not permitted.
* Women who are pregnant or nursing.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects presenting with a Crow Feet Grading score of 2 or greater for skin laxity around their periorbital area and an OSDI score of 15 or greated
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-07-25 (Actual); Primary Completion 2018-07-31 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
Skin Laxity | 5 Months
  Subjective and Objective improvement in skin laxity and wrinkles using the validation Grading Scale for Crow's Feet
  • To identify an improvement in the signs of dry eye defined as a decrease in total corneal staining after treatment compared with pre-treatment findings.

SECONDARY OUTCOMES:
Ocular Surface changes | 3 Months
  Improvement in dry eye symptoms defined by a decrease in the OSDI score by 25% and decrease in total corneal staining

CONTACTS AND LOCATIONS:
Overall Officials: Gerard D'Aversa, MD, Principal Investigator — Ophthalmic Consultants of Long Island
Locations (1):
- Ophthalmic Consultants of Long Island, Lynbrook, New York, United States

IPD SHARING:
Plan to Share IPD: No
We will not be sharing individual participant data with other researchers but do plan to present the total findings of the study.